CLINICAL TRIAL: NCT03615833
Title: Evaluation of a Strategy for Systematic Screening for Vitamin D Deficiency and Treatment in Case of Deficiency, on the Improvement of the Maximum Walking Distance in Patients With Stage 2 Lower Limb Arterial Disease.
Brief Title: Pilot Study of Vitamin D Screening Use in Peripheral Arterial Disease Patient Over Maximum Distance Walking
Acronym: First-BLINDOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-004146-41
Record Dates: First submitted 2018-07-30; First posted 2018-08-06 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral artery disease; Vitamin D
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Vitamin D deficiency (Experimental): Patients with Vitamin D deficiency, Administration of Cholecalciferol 2.5 mg (100 000 UI), once a month for 3 months
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Cholecalciferol 2.5mg (100 000 UI) , once a month for 3 months
  Other Names: Vitamin D

SUMMARY:
The prevalence of peripheral arterial disease (PAD) is greater than 15%. PAD is associated with an increased risk of cardiovascular death, coronary heart disease and stroke, with a mortality rate of 5% per year.

Most clinical evidence supports the idea that having normal vitamin D reduces cardiovascular risk. The data suggests that normalizing vitamin D levels would have a significant impact on public health, reduce costs and help control the incidence and prevalence of cardiovascular disease.

There is also a plausible physiological theory, supported by numerous observational studies, that vitamin D supplementation should be effective in improving cardiovascular outcomes, such as blood pressure, arterial stiffness, atherosclerosis, endothelial function, and clinical events.

The investigators hypothesize that routine screening for vitamin D deficiency and supplementation in case of hypovitaminosis D is effective for improving the maximum walking distance after 12 weeks of treatment in stage 2 PAD patients .

DETAILED DESCRIPTION:
At admission eligible patients are proposed to participate. Written consent is signed after complete oral and written explanation of the protocol is signed. Vitamin D level will be assessed : Patients without vitamin D deficiency will be excluded.

The influence of vitamin D supplementation on the evolution of walking distance in 12 weeks will be studied by comparing the spontaneous evolution of this walking distance, in not supplemented patients (period 1 ), and the evolution under treatment with vitamin D (period 2, afer 3 months ).

The spontaneous evolution of the walking distance will be evaluated by the difference in walking distance observed between the beginning and the end of the first Period (3 months) . The evolution of walking distance under vitamin D treatment will be evaluated by the difference in walking distance between between the beginning and the end of the second Period (3 months).

The duration of participation for a subject is equal to 6 months (2 periods of 3 months )

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting a Peripheral Arterial Disease (Stage 2)
* Affiliation to the French National healthcare system
* French speaking patients

Exclusion Criteria:

* Pregnancy
* Inability to understand the study goal
* Patients protected by decision of law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Change of the maximum walking distance on treadmill | baseline, 12 weeks and 24 weeks
  the Walking distance will be assessed during a test on a treadmill according to a standardized procedure

SECONDARY OUTCOMES:
Tolerance of vitamin D supplementation during 12 weeks of treatment (period 2) | 24 weeks
  Prevalence and description of adverse events reported by the patient in a patient book and data collected at the end of treatment
Compliance with Vitamin D supplementation | 24 weeks
  Recording of vitamin D intake by the patient in a patient booklet and counting of the number of vitamin D boxes in the V2 visit

CONTACTS AND LOCATIONS:
Overall Officials: Samir Henni, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France